CLINICAL TRIAL: NCT01625312
Title: The China PEACE (Patient-centered Evaluative Assessment of Cardiac Events) Prospective Study of Revascularization in Patients With Three-vessel Coronary Heart Disease
Brief Title: China PEACE-Prospective 3-vessel Disease Study
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Sponsor
Other Study IDs: WSGY-201202025-5
Record Dates: First submitted 2012-06-17; First posted 2012-06-21 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2014-09

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A venous blood sample of 20mL will be collected at 1-month visit and 12-month visit for biomarker analysis and storage for future genetic studies;
  A urine samples of 40mL will be collected at 1-month visit and 12-month visit for biomarker analysis and storage.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- CABG group: Three-vessel disease patients undergoing CABG at index hospitalization
- PCI group: Three-vessel disease patients undergoing PCI at index hospitalization.
- OMT group: Three-vessel disease patients undergoing no revascularization at index hospitalization

SUMMARY:
Coronary heart disease (CHD) pose a serious health threaten to population. Optimal revascularization strategy in multiple vessel coronary artery disease patients remains a subject of debate between interventional cardiologists and surgeons. Knowledge about the real-life revascularization pattern and outcomes in China is limited. By consecutively recruiting three vessel coronary heart disease patients in 25 geographically representative highest-rank hospitals, this study will examine revascularization strategy, and various real-life factors, that may affect patients lone-term recovery. Practical guidelines, appropriateness criteria and quality evaluative system for revascularization strategy will be established based on the findings, to improve patients outcomes in future finally.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a major concern in public health globally, as well as in China, and remarkable variations of resources available and health system performance have been noted. Relatively limited information is available about how evidence-based therapies are incorporated appropriately into routine clinical practice. Optimal revascularization strategy in multiple vessel coronary artery disease patients remains a subject of debate between interventional cardiologists and surgeons. Practical and applied knowledge from large unselected population is needed to guide practice and policy for quality improvement and cost reduction.

This study will enroll patients with diagnosis of three-vessel disease, or left main disease with significant lesion (over 50%) consecutively in 25 tertiary hospitals scattered all over China. At study entry, participants will be interviewed during their index hospitalization, to collect information about symptoms, functioning, quality of life, and medical care. Demographic characteristics, medical history, clinical features, diagnostic tests, medications, procedures, and in-hospital outcomes of patients will be abstracted from medical records by well trained professional abstractors. And CAG imaging will be reviewed by national and international expert panels. At 1 month, 6 month, and 12 month after discharge, participants will return to the clinic for follow up visits, a face-to-face interview will be conducted to get information about clinical events, symptoms, functioning, quality of life, and medical care during the recovery period. At 1-Month and 12-Month follow-up visit, blood and urine sample will be collected. Participants' blood samples will be stored for future biologic and genetic studies. This study will examine various real-life factors that may affect multiple vessel coronary heart disease patients recovery after PCI/CABG/medications, including patients' characteristics and treatment measures. Practical guidelines, quality evaluative system, and appropriateness criteria will be established based on the findings, to improve patients outcomes in future finally.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with diagnosis of three-vessel disease, or left main disease with significant lesion (over 50%), using selective coronary angiography at index hospitalization.

Exclusion Criteria:

* Revascularization before the index admission
* Previously enrolled in the PEACE study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In 25 tertiary hospitals with capability of Percutaneous Coronary Intervention and CABG in China, 1500 hospitalized patients diagnosed as three-vessel coronary heart disease following elective coronary angiograghy will be enrolled consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 2339 (Actual)
Dates: Start 2012-12; Primary Completion 2013-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) | 1 year
  Composite of major adverse cardiac events (MACE) including death, myocardial infarction and/or revascularization.

SECONDARY OUTCOMES:
Coronary death or myocardial infarction (fatal or non-fatal MI) | 1 year
Coronary revascularization procedure | 1 year
Presumed ischemic stroke (i.e. not known to be hemorrhagic) | 1 year
Death from all cardiovascular causes | 1 year
Re-admission | 1 year
Status of general health (SF-12) | 1 year
Quality of life (EQ-5D) | 1 year
Symptoms status (SAQ) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Jiang, M.D., Ph.D., Principal Investigator — China National Center for Cardiovascular Diseases; Harlan M Krumholz, M.D., S.M., Principal Investigator — Yale University
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Rao C, Bongiovanni T, Li X, Gao H, Zhang H, Li J, Zhao Y, Yuan X, Hua K, Hu S, Krumholz HM, Jiang L, Zheng Z; China PEACE Collaborative Group. The China Patient-Centred Evaluative Assessment of Cardiac Events (China PEACE)-Prospective Study of 3-Vessel Disease: rationale and design. BMJ Open. 2016 Feb 15;6(2):e009743. doi: 10.1136/bmjopen-2015-009743. PMID 26880670